CLINICAL TRIAL: NCT05069610
Title: A Parallel Treatment, Phase 2a, Double-blind, Randomized, Placebo-controlled, 4-arm Study to Evaluate the Safety, Tolerability, and Potential Efficacy of Intranasal AD17002 in Adult Aged 20 to 70 Years With Mild to Moderate COVID-19
Brief Title: Evaluating Safety, Tolerability, and Potential Efficacy of Intranasal AD17002 in Adults With Mild to Moderate COVID-19
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Advagene Biopharma Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AD17002-SC01
Record Dates: First submitted 2021-10-04; First posted 2021-10-06 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2021-12

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; COVID-19; Therapy, viral clearance, immunomodulator, IFN, innate
MeSH Terms: conditions — COVID-19 | interventions — heat-labile enterotoxin, E coli

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard of care + AD17002 (3 weekly doses) (Experimental): Received 3 weekly doses of AD17002 20 μg/dose of AD17002 by intranasal route
  Interventions: Biological: AD17002
- Standard of care + Placebo (3 weekly doses) (Placebo Comparator): Received 3 weekly doses of Placebo Formulation buffer by the intranasal route
  Interventions: Biological: Placebo (Formulation buffer)
- Standard of care + AD17002 (3 doses in 5 days) (Experimental): Received 3 doses of AD17002 in 5 days 20 μg/dose of AD17002 by the intranasal route on days 1, 3, and 5
  Interventions: Biological: AD17002
- Standard of care + Placebo (3 doses in 5 days) (Placebo Comparator): Received 3 doses of Placebo in 5 days Formulation buffer by the ntranasal route on days 1, 3, and 5
  Interventions: Biological: Placebo (Formulation buffer)

INTERVENTIONS:
Biological: AD17002 — A recombinant protein
  Arms: Standard of care + AD17002 (3 doses in 5 days); Standard of care + AD17002 (3 weekly doses)
Biological: Placebo (Formulation buffer) — Formulation buffer
  Arms: Standard of care + Placebo (3 doses in 5 days); Standard of care + Placebo (3 weekly doses)

SUMMARY:
AD17002 has demonstrated superior safety and efficacy as a nasal adjuvant function to an influenza vaccine in two completed clinical studies, and has innate immune modulatory and anti-inflammatory properties which could potentially be an effective treatment for SARS-CoV-2 infection.

This Phase 2a, multi-center study is set up to assess the safety, tolerability, and potential efficacy of AD17002 in participants with mild to moderate COVID-19. The Immunogenicity of repeated doses of AD17002 will also be explored.

DETAILED DESCRIPTION:
AD17002 has demonstrated superior safety and efficacy as a nasal adjuvant function to an influenza vaccine in two completed clinical studies and has innate immune-modulatory and anti-inflammatory properties which could potentially be an effective treatment for SARS-CoV-2 infection.

This Phase 2a, multi-center study is set up to assess the safety, tolerability, and potential efficacy of AD17002 in participants with mild to moderate COVID-19. The cycle threshold (Ct) was used as a surrogate biomarker for viral clearance in the exploratory study.

The COVID-19 pandemic has led to significant mortality in global populations and suppression of the economy. The prompt development of the vaccine for SARS-CoV-2 represents an unprecedented achievement for mankind, nevertheless, the unstoppable transmission of the virus highlights human's insufficient and lack of preparedness in mucosal immunity, which acts as the port of entries to not just SARS-CoV-2, but many viruses.

The AD17002, also known as LTh(αK), is an immunomodulator, which induces expression of type I and III interferons (IFN-I/III) from mucosal epithelial cells. The IFN-I/III are critical components to innate immunity, the first line defender against infection, and modulator and initiator of adaptive immunity. The IFN-I is antagonized by many SARS-CoV-2 viral proteins and studies have shown the association between IFN-I deficiency and severe COVID-19. In this study, we intended to treat subjects with AD17002, which induced nasal epithelial cells to express IFN-I/III.

Participants who meet the eligibility criteria will be isolated and confined to the study site to receive treatment for COVID-19. Eligible participants will be assigned to 2 cohorts, Cohort 1 and Cohort 2, sequentially. Cohort 1 will receive 3 doses of AD17002 or placebo weekly, while Cohort 2 will receive 3 doses of LTh(αK) or placebo every other day (Days 1, 3, and 5). Within each cohort, participants will be randomized in a 2:1 ratio to receive standard-of-care treatment and add-on therapy of AD17002 at 20 μg or placebo. Randomized participants will be assigned a participant number. The participants, site personnel, and the Sponsor will be blinded to the treatment assignment. Randomization will not be stratified and participants who withdraw from the study after starting treatment will not be replaced, except for participants who undergo sentinel dosing in Cohort 2.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 20 and ≤ 70 years
2. SARS-CoV-2 infection confirmed by real-time RT-PCR ≤ 4 days before randomization.
3. Symptoms of mild to moderate illness with COVID-19 at Screening. At least one key COVID-19 symptom should have a score of 2 or higher using the scoring system in the diary card, with the exception of fever, sense of smell, and sense of taste where participants may be enrolled with a score of 1 or higher.
4. Have a negative serum pregnancy test at Screening (for female participants of childbearing potential). A female participant who is of childbearing potential agrees to remain abstinent or use (or have their partner use) two acceptable methods of birth control within the projected duration of the study. Acceptable methods of birth control are: intrauterine device, hormonal contraception, diaphragm with spermicide, contraceptive sponge, condom, vasectomy, as per local regulations or guidelines.
5. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤ 2.5-fold of upper limit of normal (ULN) and total bilirubin ≤ 1.5-fold of ULN.
6. Creatinine clearance ≥ 50 mL/min.
7. A female participant who is not of childbearing potential is eligible without requiring the use of contraception. A female participant who is not of childbearing potential is defined as one who has either:

   1. Reached natural menopause (defined as 6 months of spontaneous amenorrhea with serum follicle-stimulating hormone levels in the postmenopausal range as determined by the laboratory, or 12 months of spontaneous amenorrhea), or
   2. At least six weeks postsurgical documented total hysterectomy and/or bilateral salpingo-oophorectomy, or
   3. Bilateral tubal ligation
8. Participant or the participant's legal representative understands the study procedures, alternative treatments available, risks involved with the study, and voluntarily agrees to participate by giving written informed consent.
9. Provide written informed consent for the study and willing to adhere to dose regimen and visit schedules.

Exclusion Criteria:

1. Participant has clinical signs suggestive of moderate (pneumonia) or more severe illnesses with COVID-19 (as defined in the Taiwan CDC "Interim Guideline for Clinical Management of SARS-CoV-2 Infection Version 13" (Taiwan CDC, Clinical Management of SARS-CoV-2 Infection).
2. Participation in any other clinical study of an investigational agent treatment for SARS- CoV-2 infection within 30 days prior to the first IMP dosing.
3. Participant who has a history of confirmed SARS-CoV-2 infection.
4. Concurrent treatment with other agents with actual or possible direct acting antiviral activity against SARS-CoV-2 < 24 hours prior to the first IMP dosing.
5. History of severe renal disease (treatment with dialysis or phosphate binders) or clinically apparent hepatic impairment (e.g., jaundice, cholestasis, hepatic synthetic impairment, active hepatitis).
6. Impaired cardiac function or clinically significant cardiac diseases as judged by the Investigator.
7. History of anaphylaxis reaction to any known or unknown cause.
8. Immunosuppressed persons as result of illness (e.g., HIV infection) or treatment.
9. Documented history of Bell's palsy.
10. History of allergic reaction to kanamycin.
11. Immunosuppressive treatment within 3 months prior to the Screening Visit.
12. Ongoing treatment with any specific immunotherapy at the time of the Screening Visit.
13. Assessed by the Investigator to be ineligible to participate in the study.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-12-18 (Actual)

PRIMARY OUTCOMES:
The proportion of participants who experience adverse events | 7 weeks
  Clinicians and Patients reported AEs in the study period (7 weeks)
The proportion of participants with treatment-emergent adverse events (TEAE) leading to investigational medicinal products (IMPs) discontinuation | 7 weeks
  Measuring and recording the AEs caused by treatment.
The nasal tolerability to investigational medicinal products (IMPs) | 7 weeks
  Nasal symptoms will be assessed by participants and ear-nose-throat (ENT) specialists on symptoms include runny nose, stuffy nose, nasal discomfort, sneezing, lacrimation, change in vision, red eyes, facial swelling, nasal pain.
  Symptom Score Guide: 0= None; 1= Mild; 2= Moderately; 3= Severe

SECONDARY OUTCOMES:
The time to proportions of participants have a Ct≥30 | 7 weeks
  Measuring the RT-PCR on RdRp and E gene
Time to recovery* of fever (days) | 7 weeks
  Fever is defined as temperatures of ≥ 36.6°C (axilla), or ≥ 37.2°C (oral), or ≥ 37.8°C (rectal or tympanic) over a 48-hour period. Recovery of fever is defined as occurring when body temperature is < 36.6°C (axilla), or < 37.2°C (oral), or < 37.8°C (rectal or tympanic) over a 48-hour period.
Time to recovery* of sore throat (days) | 7 weeks
  Recovery of sore throat is defined as occurring when the symptom of sore throat has resolved to a score of 0 over a 48 hour period
Time to recovery* of cough (days | 7 weeks
  Recovery of cough is defined as occurring when the symptom of cough has resolved to a score of 0 over a 48 hour period
Time to recovery* of fatigue (days). | 7 weeks
  Recovery of fatigue is defined as occurring when the symptom of fatigue has resolved to a score of 0 over a 48 hour period
Time to recovery* of muscle/body pain (days) | 7 weeks
  Recovery of muscle/body pain is defined as occurring when the symptom of muscle/body pain has resolved to a score of 0 over a 48 hour period
Time to recovery* of other symptoms (days) | 7 weeks
  Recovery of symptom is defined as occurring when the symptom has resolved to a score of 0 over a 48 hour period
The mean change from baseline to each specified time point on National Early Warning Score 2 (NEWS2) | 7 weeks
  Clinicians or study staffs report the NEWS 2 scores for each subject.

OTHER OUTCOMES:
Changes to anti-SARS CoV-2 antibody titers from baseline | 7 weeks
  Measuring virus-specific IgG within serum
Changes to pre-specified immunological markers | 7 weeks
  Measuring the IL6, lymphocyte count and neutrophil-to-lymphocyte ratio.
Viral genome integrity analysis | Cohort 1, 3 weeks; Coohort 2, 8 days
  Measuring the ratio of different viral gene expressed after treatments

CONTACTS AND LOCATIONS:
Overall Officials: Mingi Chang, PhD, Study Director — Advagene Biopharma
Locations (2):
- Taiwan (2):
  - Advagene Biopharma, Taipei
  - Chang Gun Medical Foundation, Taoyuan District

IPD SHARING:
Plan to Share IPD: No